CLINICAL TRIAL: NCT00000794
Title: Phase II Randomized Open-Label Trial of Atovaquone Plus Pyrimethamine and Atovaquone Plus Sulfadiazine for the Treatment of Acute Toxoplasmic Encephalitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 237; ANRS 039; 11214 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Toxoplasmosis, Cerebral; HIV Infections
Keywords: Pyrimethamine; Leucovorin; Drug Therapy, Combination; Encephalitis; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents; Clarithromycin; atovaquone; Toxoplasmosis, Cerebral; Sulfadiazine
MeSH Terms: conditions — Toxoplasmosis, Cerebral; HIV Infections; Encephalitis; Acquired Immunodeficiency Syndrome | interventions — Sulfadiazine; Clarithromycin; Atovaquone; Pyrimethamine; Leucovorin

INTERVENTIONS:
Drug: Sulfadiazine
Drug: Clarithromycin
Drug: Atovaquone
Drug: Pyrimethamine
Drug: Leucovorin calcium

SUMMARY:
To evaluate the efficacy, safety, and tolerance of atovaquone with either pyrimethamine or sulfadiazine in AIDS patients with toxoplasmic encephalitis.

AIDS patients with toxoplasmic encephalitis who receive the standard therapy combination of sulfadiazine and pyrimethamine experience a high frequency of severe toxicity. Atovaquone, an antibiotic that has demonstrated efficacy against toxoplasmosis in animal models and in preclinical testing has been well tolerated, is now available as a suspension, which is more readily absorbed than the tablet form of the drug. The efficacy and safety of atovaquone in combination with sulfadiazine or pyrimethamine will be studied.

DETAILED DESCRIPTION:
AIDS patients with toxoplasmic encephalitis who receive the standard therapy combination of sulfadiazine and pyrimethamine experience a high frequency of severe toxicity. Atovaquone, an antibiotic that has demonstrated efficacy against toxoplasmosis in animal models and in preclinical testing has been well tolerated, is now available as a suspension, which is more readily absorbed than the tablet form of the drug. The efficacy and safety of atovaquone in combination with sulfadiazine or pyrimethamine will be studied.

Seventy patients are randomized to receive atovaquone with either pyrimethamine or sulfonamides for up to 48 weeks. Additionally, three cohorts of 10 patients each who have a history of treatment-limiting toxicity to pyrimethamine, sulfadiazine, or both drugs receive atovaquone plus the alternate drug or atovaquone plus clarithromycin. All patients receiving pyrimethamine also receive leucovorin protection.

PER AMENDMENT 4/3/96:

The open treatment groups are: Atovaquone plus pyrimethamine for patients with acute toxoplasmic encephalitis who have no treatment limiting toxicity to pyrimethamine, and Atovaquone plus clarithromycin for patients with acute toxoplasmic encephalitis who have treatment limiting toxicity to both pyrimethamine and sulfadiazine. The following arms closed on 12/22/95: Randomization to the atovaquone plus sulfadiazine arm for patients with acute toxoplasmic encephalitis who had no treatment limiting toxicity to pyrimethamine or sulfonamides, and Atovaquone plus sulfadiazine for patients with acute toxoplasmic encephalitis who had treatment limiting toxicity to pyrimethamine. The following arm closed on 9/26/95: Atovaquone plus pyrimethamine for patients with acute toxoplasmic encephalitis who had treatment limiting toxicity to sulfonamides. NOTE: Any patients enrolled in previous versions will continue to be treated with that same drug treatment and followed under their previous version guidelines.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine for PCP prophylaxis.

PER AMENDMENT 4/3/96:

* History of treatment limiting toxicity to pyrimethamine. Patients with a history of treatment limiting toxicity to both pyrimethamine and sulfonamides will be assigned to receive atovaquone plus clarithromycin.

Patients must have:

* Documented HIV infection or diagnosis of AIDS (except for CD4 count < 200 cells/mm3).
* Toxoplasmic encephalitis.
* Ability to give informed consent or legal designee who could give consent.

PER AMENDMENT 4/3/96:

* NOTE - A history of treatment limiting toxicity to both pyrimethamine and sulfonamides will result in the patient being enrolled in the atovaquone plus clarithromycin arm.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Coma.
* Opportunistic infection that requires either acute or maintenance treatment with disallowed medications.
* Any infections or neoplasms of the central nervous system other than Toxoplasma, HIV encephalopathy, or syphilis.
* Unable to take oral study drugs.
* Malabsorption (i.e., three or more episodes of diarrhea per day that has caused >= 10 percent loss of body weight over the past 4 weeks).
* Positive CSF or serum for Cryptococcus antigen or culture (a positive serum antigen only is acceptable, provided patient received prior antifungal therapy and is on maintenance, and the likelihood of recurrence is low).
* Malignancy requiring use of cytotoxic chemotherapy.
* Medical or social condition that would adversely affect study participation or compliance.

Concurrent Medication:

Excluded:

* Trimethoprim-sulfamethoxazole.
* Primaquine.
* Sulfonamides.
* Antifolates.
* Dapsone.
* Clarithromycin (except for patients in the cohort to receive this drug).
* Azithromycin.
* Clindamycin.
* Other macrolides.
* Gamma interferon.
* Metoclopramide.
* G-CSF or GM-CSF.

Excluded in patients receiving clarithromycin as study drug:

* Terfenadine, astemizole, or any other long-acting, non-sedating antihistamines.

PER AMENDMENT 4/3/96:

* Cisapride - may increase GI motility and may increase drug absorption.

Patients with the following prior conditions are excluded:

* History of treatment-limiting toxicity to atovaquone.
* Receipt of > 96 hours (per amendment) of treatment prior to study entry for the current episode of toxoplasmic encephalitis.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luft B, Study Chair; Chirgwin K, Study Chair
Locations (16):
- United States (16):
  - USC CRS, Los Angeles, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio

REFERENCES:
- [Background] Chirgwin K, Hafner R, Leport C, Remington J, Andersen J, Bosler EM, Roque C, Rajicic N, McAuliffe V, Morlat P, Jayaweera DT, Vilde JL, Luft BJ. Randomized phase II trial of atovaquone with pyrimethamine or sulfadiazine for treatment of toxoplasmic encephalitis in patients with acquired immunodeficiency syndrome: ACTG 237/ANRS 039 Study. AIDS Clinical Trials Group 237/Agence Nationale de Recherche sur le SIDA, Essai 039. Clin Infect Dis. 2002 May 1;34(9):1243-50. doi: 10.1086/339551. PMID 11941551